| Official Title: |
|------------------------------------------------------------------|
| Tailoring the Chicago Parent Program for the Foster Care Setting |
| Identifier: |
| NCT05856435 |
| Document: |
| Informed Consent Form – Participant Permission |

CCH IRB Approval Date: 10/12/2023 IRB Number: 2022-0228

**Title of research study:** Adapting Chicago Parent Program for Foster Care – Pilot Study

## **Key Information:**

The following is a short summary of this study to help you decide whether to be a participant in it. More detailed information about the study is listed later in this form. This document does not replace the discussion you should have with the research team about this study including having any questions or concerns answered.

This is a consent form. It explains this research study. If you decide that you want to be in this research study, then you will sign this form to show that you agree to be part of this study. If you sign this form, you will receive a signed copy of it for your records.

## Reason for the study:

The main reason for this research study is to adapt and pilot the Chicago Parent Program (CPP) for foster caregivers (CPP-FC). CPP uses 12 sessions to deliver content. Topics include concepts such as the value of child-centered time; family routines and traditions; use of praise and encouragement; use of rewards for challenging behavior; limit setting; following through on commands; use of behavior management strategies such as ignoring, distraction, and time-out; managing stress; and problem-solving. Facilitators use video vignettes, handouts, and role-play during the sessions to support content delivery and engage parents in the material.

You are being asked to participate in this study because you are a licensed foster caregiver or a kinship caregiver to a child in foster care between the ages of 2 and 8 years old who has been placed in your home within the past 45 days.

#### **Procedures:**

We expect that you will be in this research study for approximately 3 months.

After signing this consent form, you will be asked to complete electronic surveys about the amount of stress that you experience as a caregiver to a child in foster care, your level of confidence in managing the behaviors of your foster child, and an inventory of the behaviors of your foster child. The survey will also ask you some questions about yourself, such as your age, gender, race and ethnicity, education, household structure and income, and your length of experience as a foster or kinship caregiver.

You will be asked to attend a total of 12 sessions of the Chicago Parent Program adapted for foster caregivers (CPP-FC). The first 11 sessions occur weekly, and the final CPP-FC session occurs 4 weeks after the 11<sup>th</sup> session. All sessions will take place virtually using Microsoft Teams, and all sessions will be recorded. Each session will last

### **Investigator:**

Sarah Beal, PhD

## **Contact Info:**

Meera Patel, Study Coordinator

Meera.Patel@cchmc.org

# **CCHMC Protocol #:**

2022-0228

#### **Intervention Name:**

Chicago Parent Program Adapted for Foster Care (CPP-FC)

**Funding**: National Institutes of Health

CCH IRB Approval Date: 10/12/2023 IRB Number: 2022-0228

approximately 2 hours. After each session, you will be asked to complete homework assignments and electronic surveys to give feedback based on that week's program content.

After the final CPP-FC session, you will repeat the baseline electronic surveys on the amount of stress that you experience as a caregiver to a child in foster care, your level of confidence in managing the behaviors of your foster child, and an inventory of the behaviors of your foster child. There will be additional electronic surveys on your overall satisfaction with the CPP-FC program. If your foster child has changed placements during the study, you will not complete surveys on child behavior at this session. We will also ask you to take part in a semi-structured interview with the researchers and give feedback about the program, and you will be given the opportunity to suggest ways that we can improve CPP-FC. If you have multiple caregivers in your household who participate in CPP-FC sessions, all caregivers in your household will be invited to participate in the interview. This interview will take approximately 45 minutes to complete and will be conducted virtually via Microsoft Teams. These interviews will be recorded.

More detailed information about the study procedures can be found under "(Detailed Procedures)"

### Risks to Participate:

This study is deemed minimal risk. The only potential risk is a loss of confidentiality, and the research team has multiple systems in place to ensure that your information stays private.

### Benefits to Participate:

We cannot promise any benefits to you or others from your taking part in this research. However, possible benefits include an increased knowledge on how to manage the behaviors of your foster child(ren). If you are a licensed caregiver, you may also be eligible to receive ongoing training hours through your licensing agency.

#### Other Options:

Participation in research is completely voluntary. Your decision to participate or not to participate will not affect the care you or your foster child receive at Cincinnati Children's Hospital.

Your alternative to participating in this research study is to not participate.

## Cost to Participate:

Participating in this study will not cost you anything.

#### Payment:

If you agree to take part in this research study, we will pay you up to \$155.

CCH IRB Approval Date: 10/12/2023 IRB Number: 2022-0228

- Baseline surveys \$10
- Weekly CPP homework and feedback- \$5 (\$5 x 11 weekly sessions)
- Weekly CPP session attendance \$5 (\$5 x 11 weekly sessions)
- End of program surveys- \$15
- End of program semi-structured interview- \$20 (per household)
  - o If the interview takes more than 60 minutes to complete, you will receive an additional \$10, making your total possible compensation \$165.

## **Additional Study Information:**

The following is more detailed information about this study in addition to the Key Information.

## If I have Questions or would like to know about:

| ? Who to talk to | You can call | ₿ At |
|---|---|---|
| <ul> <li>Emergencies</li> <li>General study questions</li> <li>Any research concerns or complaints</li> </ul> | Sarah Beal, PhD | Phone: (513) 636-4614 |
| <ul> <li>Emergencies</li> <li>General study questions</li> <li>Any research concerns or complaints</li> </ul> | Meera Patel Lead Study Coordinator | Phone: (513) 803-1674 |
| <ul> <li>Your rights as a research participant</li> </ul> | Institutional Review Board This is a group of scientists and community members who make sure research meets legal and ethical standards. | Phone: (513) 636-8039 |

#### **Detailed Procedures:**

At the baseline study timepoint, you will provide informed consent, and complete surveys about:

- The amount of stress that you experience as a caregiver to a child in foster care
- Your level of confidence in managing the behaviors of your foster child
- An inventory of the behaviors of your foster child.

CCH IRB Approval Date: 10/12/2023 IRB Number: 2022-0228

• The survey will also ask you some questions about yourself, such as your age, gender, race and ethnicity, education, household structure and income, and your length of experience as a foster or kinship caregiver.

Sessions 1 – 11 of the CPP-FC program will occur on a weekly basis. Sessions will be conducted virtually via Microsoft Teams by two trained CPP-FC program facilitators. There will be 5-7 other foster or kinship caregivers participating in these sessions with you. Each session will last approximately 2 hours, and all sessions will be recorded. Activities during sessions involve:

- Video vignettes on managing child behaviors
- Role-plays on how to manage child behaviors
- Group discussions based on that week's program content

After each session, you will be asked to complete:

- Weekly homework assignments based on that week's program content
- A survey on your level of satisfaction with weekly program content

The final CPP-FC session will occur 4 weeks after the 11<sup>th</sup> session. After the final session, you will be asked to complete surveys about:

- The amount of stress that you experience as a caregiver to a child in foster care
- Your level of confidence in managing the behaviors of your foster child
- An inventory of the behaviors of your foster child.
- Your overall satisfaction on the CPP-FC program.

We will also ask you to participate in a semi-structured interview with the research team about your satisfaction with CPP-FC content, and you will be given the opportunity to provide feedback on how we can improve CPP-FC. If multiple caregivers from your household participate in CPP-FC sessions, they will also be invited to participate in the interview.

## Change of Mind/Study Withdrawal:

You can leave the research at any time; it will not be held against you.

If you decide to leave the research, contact the investigator or the study coordinator in writing (a mailed letter or an email) so they can withdraw you from the study.

### Privacy:

Efforts will be made to limit the use and disclosure of your personal information, including research study records, to people who have a need to review this information.

CCH IRB Approval Date: 10/12/2023 IRB Number: 2022-0228

We cannot promise complete privacy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization. This study uses HIPAA-compliant software such as Microsoft Teams for conducting recorded CPP-FC sessions and interviews, and all study files are kept on password-protected computers on secure CCHMC servers via HIPAA-compliant hard drives and electronic file storage systems, such as Microsoft OneDrive and REDCap.

Data collected for or generated from this study could be shared and used for future research. Data may be shared with other collaborators at Cincinnati Children's and possibly with outside collaborators, who may be at another institution or for-profit company.

If information that could identify you is removed from your information collected during this research, that information could be stored and used for future research studies or distributed to another investigator for future research studies without your additional informed consent.

#### **SIGNATURES**

The research team has discussed this study with you and answered all of your questions. Like any research, the researchers cannot predict exactly what will happen. Once you have had enough time to consider whether you should participate in this research, you will document your permission by signature below.

| Printed Name of Research Participant | - | |
|---------------------------------------------------------|------|---|
| Signature of Research Participant<br>Indicating Consent | Date | _ |
| Signature of Individual Obtaining Consent | | |

You will receive a copy of this signed document for your records.